CLINICAL TRIAL: NCT03725046
Title: Evaluation of the Impact of an Optimized Communication Between Hospital and Community on the Readmission at the Emergency Department for an Adverse Drug Event : Randomized Controlled Trial
Brief Title: Impact of an Optimized Communication on the Readmission for Adverse Drug Event
Acronym: URGEIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UF7591
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-11

CONDITIONS: Adverse Drug Event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual information transmission after ED admission (No Intervention): The emergency department (ED) sends to the referring doctor a letter to inform him about the reason of consultations in the emergency department (mail currently realized as part of the care process).
- Optimized information transmission after ED admission (Experimental): Sending to the community referring physician by the emergency department an discharge report containing the reason for emergency consultations (report currently made as part of the treatment). Within 72 hours (working hours), the Emergency Clinical Pharmacist contacts the referring physician and the patient's community pharmacist to discuss how to manage the ADE. In parallel, a second report, summary of the ADE (ADE-report), is sent to them. The ADE-report, written and validated by the investigators (emergency physician and clinical pharmacist), includes the type of ADE, the suspected drug(s) and other recommendations: therapeutic modification, referral to specialized consultations (geriatrics ...).
  Interventions: Other: Optimized information transmission

INTERVENTIONS:
Other: Optimized information transmission — Sending to the community referring physician by the emergency department an discharge report containing the reason for emergency consultations (report currently made as part of the treatment). Within 72 hours (working hours), the Emergency Clinical Pharmacist contacts the referring physician and the patient's community pharmacist to discuss how to manage the ADE. In parallel, a second report, summary of the ADE (ADE-report), is sent to them. The ADE-report, written and validated by the investigators (emergency physician and clinical pharmacist), includes the type of ADE, the suspected drug(s) and other recommendations: therapeutic modification, referral to specialized consultations (geriatrics ...).
  Arms: Optimized information transmission after ED admission

SUMMARY:
Emergency departments (EDs) are a crucial element of health care systems as they constitute the interface between hospital and communities. The goals of the ED are to make an initial diagnosis and deliver urgent and critical care 24 hours per day and 365 days a year. Also, many Adverse Drug Events (ADEs) are not identified by emergency physicians. ADEs are injuries resulting from a drug related medical intervention. Their detection, documentation and reporting are essential for adequate medical care and knowledge of risk/benefit profiles of medication throughout their lifecycle. However, a number of studies indicate that in clinical practice the under-reporting of ADEs is a pervasive and widespread problem. The main reasons for under-reporting were difficulty in determining the cause of the ADE, lack of time, poor integration of ADE-reporting systems and uncertainty about reporting procedures. Successful treatment of ADEs depends on the ability of physicians to attribute ADEs to a medication. Some studies have reported that not only pharmacists but also pharmacy student were one of the best health care providers to establish medication history and detected ADEs.

It has also been shown that a clinical pharmacist, within the emergency medical team, can improve the detection of ADE through drug expertise and reliable drug history. This approach has been adopted at Montpellier University Hospital since November 2011. During the initial diagnosis of the ADE, the revision of a drug treatment at risk cannot be carried out in emergency department by the emergency physician. Indeed, the latter intervenes punctually but he is not the patient's referring doctor. Guidance and follow-up of the patient throughout the care journey is the responsibility of the referring physician, sometimes accompanied by the pharmacist. It is therefore very important that a relevant information detected at the hospital can be passed on to the referring health professionals who will review and adapt the treatment. The city-hospital link is essential to guarantee the continuity and the consistence of the care process. When a patient is discharging with the emergency department, the outgoing mail often mentions only the reason for admission, and the information concerning the detection or suspicion of an ADE is not systematically stipulated. However, this information is essential to trigger a process of therapeutic revision (therapeutic modification, therapeutic education, referral to specialized consultations ...) that will prevent the recurrence of the ADE and therefore the readmission to emergency department. To date, the rate of readmission to emergency department after a first visit related to an ADE is between 3.6 and 18.7%.

Our goal is to evaluate the impact at 6 months of a medical-pharmaceutical follow-up and the optimization of the city-hospital link following an admission at emergency department for ADE, on the readmission to emergency department for the same ADE.

This is a single-center randomized, controlled, open-label, two-arm, parallel, "usual information transmission" or "optimized information transmission" study. The duration of a patient's follow-up is 6 months.

Each patient with an occurring ADE detected during emergency department admission could be participating in the study.

Specific management of the experimental group: Sending to the community referring physician by the emergency department an discharge report containing the reason for emergency consultations (report currently made as part of the treatment). Within 72 hours (working hours), the Emergency Clinical Pharmacist contacts the referring physician and the patient's community pharmacist to discuss how to manage the ADE. In parallel, a second report, summary of the ADE (ADE-report), is sent to them. The ADE-report, written and validated by the investigators (emergency physician and clinical pharmacist), includes the type of ADE, the suspected drug(s) and other recommendations: therapeutic modification, referral to specialized consultations (geriatrics ...)

Control group: The emergency department sends to the referring doctor a letter to inform him about the reason of consultations in the emergency department (mail currently realized as part of the care process).

Primary outcome measure: Percentage of patients who had at least one readmission for the same reason in the emergency department within 6 months of the initial exit. This information will be collected during a telephone call with the patient and the referring physician.

ELIGIBILITY:
Inclusion criteria:

* Patient over 18 years old
* Patient to whom an ADE is detected
* Possibility of carrying out a pharmaceutical consultation/interview
* Patient who has consented to participate
* Patient affiliated to the social welfare policy
* Patient who declared a referent medical doctor

Exclusion criteria:

* ADE linked to an emergency care activity
* Voluntary medical intoxication
* Impossibility of recovering the patient's drug history
* Under 18
* Pregnancy
* Participating in another category 1 interventional drug study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who had at least one readmission in the emergency department for the same reason | within 6 month of the initial visit

SECONDARY OUTCOMES:
Percentage of patients who had at least one readmission in the emergency department for any reason | within 6 month of the initial visit
Percentage of patients hospitalized for ADE at least once | within 6 month of the initial visit
Percentage of patients hospitalized for any reason at least once | within 6 months of the initial visit
Potentially avoidable hospitalization rate | 6 months
Mortality rate related to ADE and all other causes | 6 months
Number of medical consultations with a general community practitioner in connection with ADE and all causes combined | 6 months
Number of medical consultations with a specialist community practitioner in connection with ADE and all causes combined | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maxime VILLIET, PharmD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villiet M, Laureau M, Perier D, Pinzani V, Giraud I, Lohan L, Bobbia X, Mercier G, Jaussent A, Macioce V, Sebbane M, Faucanie M, Breuker C. Emergency Department Visits for Medication-Related Events With vs Without Pharmacist Intervention: The URGEIM Randomized Clinical Trial. JAMA Intern Med. 2025 Jun 1;185(6):669-678. doi: 10.1001/jamainternmed.2025.0640. PMID 40293767
- [Derived] Breuker C, Faucanie M, Laureau M, Perier D, Pinzani V, Marin G, Sebbane M, Villiet M. Impact of a medico-pharmaceutical follow-up and an optimized communication between hospital and community on the readmission to the emergency department for an adverse drug event: URGEIM, study protocol for a randomized controlled trial. Trials. 2021 Aug 6;22(1):521. doi: 10.1186/s13063-021-05501-4. PMID 34362410